CLINICAL TRIAL: NCT04825912
Title: Resilience Measurement, Prediction, and Its Role in Older Adults With Late-Stage Lung Cancer
Brief Title: Resilience Measurement in Older Adults With Late-Stage Lung Cancer
Acronym: SST Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00106533
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer Stage III; Lung Cancer Stage IV
MeSH Terms: conditions — Lung Neoplasms | interventions — Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Advanced Lung Cancer (Experimental): Older adults with stage III or stage IV lung cancer will be enrolled in the Self-System Therapy intervention to treat illness-related distress, depression, and to enhance self-efficacy via delivery of behavioral coping skills across a period of 10 weeks.
  Interventions: Behavioral: Self System Therapy for Older Adults with Advanced Lung Cancer (SST-LC) Resilience

INTERVENTIONS:
Behavioral: Self System Therapy for Older Adults with Advanced Lung Cancer (SST-LC) Resilience — The SST-LC is a brief structured intervention deliverable by video conference. The SST-LC Resilience protocol will incorporate behavioral strategies designed to meet the needs of older adults with lung cancer, including examining individual and shared expectations for lung cancer care, identifying discrepancies between expectations and realistic possibilities, and modifying stress-exacerbating behaviors. The focus will be to test measures of resilience during the intervention period.

SUMMARY:
The purpose of this study to test measures of physical and psychological resilience while using Self-System therapy (SST), to treat depression and lung-cancer-related distress in older adults (65 years and older).

DETAILED DESCRIPTION:
The investigator will examine the feasibility of delivering measures of psychological and physical resilience while delivering the SST intervention. The investigator will also examine whether participation in SST can help alleviate symptoms of depression and distress while helping improve overall physical functioning in older adults with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* English-speaking
* The patient has a diagnosis of late-stage (III-IV) lung cancer and is living at his/her home.

Exclusion Criteria:

* Unable to provide informed consent
* Visual or hearing impairments that preclude participation
* Serious mental illness

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ramos, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adults With Advanced Lung Cancer
Started | 18
Completed | 14
Not Completed | 4
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (3.976)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Confidence in Behavior as Measured by the Cancer Behavior Inventory
Description: The Cancer Behavior Inventory measure will be used for rating confidence in behavior. The measure consist of 12 items. Scores range from 12-108 with higher scores indicating greater confidence.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 80.89 (21.13)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 85.92 (13.97)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 93.23 (11.19)

2. Secondary Outcome: Coping Skills Related to Stress as Measured by the Brief COPE (Coping Orientation to Problems Experienced)
Description: The Brief COPE measure will be used for rating coping skills related to stress. The measure consists of 28 items. Scores range from 28-112 with higher scores indicating lower stress.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 55.72 (10.29)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 58.54 (11.70)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 57.62 (14.23)

3. Secondary Outcome: Resilience as Measured by the CD-RISC-25 (Connor-Davidson Resilience Scale)
Description: The CD-RISC-25 will be used for measuring resilience. The measure consists of 25 items with a scaling of 0-4. Scores range from 0-100, with higher scores being an indicator of higher resilience.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 73.16 (15.06)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 75.69 (7.67)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 78.00 (9.65)

4. Secondary Outcome: Depression as Measured by the Beck Depression Inventory (BDI-II)
Description: Depression will be measured using the Beck Depression Inventory (BDI-II). The measure consists of 21 items. The BDIII is scored by summing the ratings for the 21 items. Each item is rated on a 4-point scale ranging from 0 to 3 with a total score range of 0 to 63. Higher scores indicate greater depression.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 9.06 (4.56)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 7.92 (5.09)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 8.23 (4.38)

5. Secondary Outcome: Positive Affect as Measured by the PANAS (Positive and Negative Scale)
Description: The PANAS measure will be used for rating to measure positive affect. Scores range from 10-50, with higher scores indicating higher positive affect.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 32.72 (8.38)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 34.61 (9.49)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 36.15 (7.20)

6. Secondary Outcome: Negative Affect as Measured by the PANAS (Positive and Negative Scale)
Description: The PANAS measure will be used for rating to measure negative affect. Scores range from 10-50, with higher scores indicating higher negative affect.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 18.04 (15.44)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 17.31 (5.60)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 17.54 (7.80)

7. Secondary Outcome: Physical Activity as Measured by the PASE (Physical Activity Scale for the Elderly)
Description: Physical Activity will be measured using the Physical Activity Scale for the Elderly (PASE). The instrument is comprised of 12 self-reported occupational, household and leisure activities items over a one-week period. The total PASE score is computed by multiplying either the time spent in each activity (hours per week) or participation (i.e., yes/no) in an activity, by empirically derived item weights and then summing overall activities. The PASE instrument uses frequency, duration, and intensity level of activity over the previous week to assign a score. The overall PASE score ranges from 0 to 793, where a higher score indicates more physical activity.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected on 5 participants at 8 weeks or at 10 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
score on a scale
  Baseline | 101.06 (76.24)
  8 weeks: number analyzed (Participants) | 13
  8 weeks | 110.23 (82.14)
  10 weeks: number analyzed (Participants) | 13
  10 weeks | 109.17 (73.50)

8. Secondary Outcome: Pain Interference as Measured by the PROMIS PI (Patient-Reported Outcomes Measurement Information System Pain Interference)
Description: The Pain Interference PROMIS Scale measure will be used for rating pain interference in daily living. The measure consists of 6 items. Scores range from 6-30, with higher scores indicating higher pain interference.
Time Frame: Baseline, 8 weeks, 10 weeks
Population: Data not collected.
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants Who Completed the QUALE (Quality of Life at the End of Life)
Description: The Quality-of-Life measure consists of 26 items. Scores range from 26-130, with higher scores indicating higher quality of life. The measure will be offered to assess how many total participants complete the measure in its entirety.
Time Frame: Baseline, 8 weeks, 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adults With Advanced Lung Cancer
Number analyzed (Participants) | 18
Participants
  Baseline | 18
  8 weeks | 13
  10 weeks | 13

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Arm/Group | Adults With Advanced Lung Cancer
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-05-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT04825912/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT04825912/ICF_000.pdf